CLINICAL TRIAL: NCT00123422
Title: Innovation Methods to Augment Pulmonary Rehabilitation
Brief Title: Innovation in Pulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F3845-R
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Pulmonary Disease; Pulmonary Emphysema
Keywords: Breathing exercise; Exercise Therapy; Helium; Oxygen inhalation therapy; Pulmonary emphysema; Pulmonary ventilation; Rehabilitation
MeSH Terms: conditions — Lung Diseases; Pulmonary Emphysema | interventions — heliox; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Breathing retraining (Experimental): Exercise training with computerized training program
  Interventions: Behavioral: Breathing retraining
- Heliox (Experimental): Exercise training with helium oxygen combination
  Interventions: Behavioral: Heliox
- Exercise (Active Comparator): Exercise training
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Breathing retraining — exercise training with computerized training program
  Arms: Breathing retraining
Behavioral: Heliox — exercise training with a helium oxygen combination
  Arms: Heliox
Behavioral: Exercise — exercise training
  Arms: Exercise

SUMMARY:
The purpose of this study was to compare the effect of exercise treatment combined with breathing retraining (a computerized feedback program), with exercise treatment combined with heliox (a helium and oxygen combination), with exercise only in patients with moderate to severe chronic obstructive pulmonary disease. This was an 8-week intervention study.

DETAILED DESCRIPTION:
Dynamic hyperinflation limits exercise tolerance in patients with chronic obstructive pulmonary disease (COPD). Recently, several innovative approaches have been developed to reduce the burden of dynamic hyperinflation. Two such innovations, ventilation-feedback training and Heliox supplementation during exercise show great promise and posit a reduction in dynamic hyperinflation as a key to their effectiveness. In our recently completed trial, when age, FEV1 and RV/TLC were controlled, exercise plus VF (E+VF) was superior to E training alone (E only) or VF training alone in improving exercise tolerance. The mechanism responsible for this difference was, in part, a reduction in exercise-induced dynamic hyperinflation secondary to a change in breathing pattern. In additional preliminary studies, we determined that exercise tolerance can be increased when patients exercise while inhaling Heliox. Similar to VF, the mechanism for exercise improvement with Heliox was a reduction in exercise-induced dynamic hyperinflation. Although both interventions are promising, there are no definitive data to support use of either intervention as a standard of care for pulmonary rehabilitation.

Hypothesis/Research Questions Overview: The two primary hypotheses are that patients with moderate-severe COPD who successfully complete eight weeks of (a) E+VF training will achieve longer exercise duration than patients randomly assigned to E only and (b) E+heliox training will achieve longer exercise duration than patients randomly assigned to E only.

Methods: This study was a randomized controlled clinical trial. After baseline testing is completed, 103 subjects with moderate-severe COPD were randomized into one of three groups: E+VF, E+Heliox and E training only. Follow-up testing was completed at 8 weeks. testing, activity monitoring, and dyspnea measurements. After baseline testing was completed, randomized subjects trained in the Physical Performance Laboratory three times weekly. Exercise prescriptions were standardized and based on data from the exercise stress test.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age
* FEV1 70%
* FEV1/FVC <70%
* RV/TLC > 120%

Exclusion Criteria:

* Respiratory infection/exacerbation within last 4 weeks
* Exercise limiting heart disease
* Primary asthma
* Congestive heart failure New York Heart Association (NYHA) Class III-IV
* Exercise limiting peripheral arterial disease or arthritis
* Inability to walk on a treadmill

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2005-10; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen G. Collins, PhD RN, Principal Investigator — Edward Hines Jr. VA Hospital
Locations (1):
- Edward Hines, Jr. VA Hospital, Hines, Illinois, United States

REFERENCES:
- [Result] Collins EG, Jelinek C, O'Connell S, Butler J, McBurney C, Gozali C, Reda D, Laghi F. Contrasting breathing retraining and helium-oxygen during pulmonary rehabilitation in COPD: a randomized clinical trial. Respir Med. 2014 Feb;108(2):297-306. doi: 10.1016/j.rmed.2013.10.023. Epub 2013 Nov 5. PMID 24238770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 192 patients were screened for eligibility in the study. 103 patients were randomly assigned to the one of the 3 groups. Patients were not randomized for the following reasons: PFT did not qualify (n=47), cardiac problems (n=13), changed mind (n=9), non-compliant (n=6), time constraints (n=5), too debilitated (n=3), other (n=6).
Period: Overall Study
Arm/Group | Breathing Retraining | Heliox | Exercise
Started | 35 | 33 | 35
8-week Testing | 32 | 30 | 27
Completed | 31 | 27 | 25
Not Completed | 4 | 6 | 10
Not completed — Physician Decision | 2 | 2 | 6
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — Lost to Follow-up | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Breathing Retraining | Heliox | Exercise | Total
Number analyzed (Participants) | 35 | 33 | 35 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (10) | 70 (9) | 69 (7) | 69 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 33 | 31 | 34 | 98
Region of Enrollment [Number; unit: participants]
  United States | 35 | 33 | 35 | 103
Smoking history [Mean (Standard Deviation); unit: pack/years] — Smoking history was measured in pack/years. This is the number of packs of cigarettes smoked per day multiplied by the number of years of smoking.
  pack/years | 62 (37) | 67 (40) | 68 (48) | 64 (42)
FEV1 percent predicted [Mean (Standard Deviation); unit: percent] — The FEV1 (forced expiratory volume in 1 second) is a measure of pulmonary function. It is the amount of air that a person can blow out in one second. This value is reported as the percentage of predicted normal.
  percent | 45 (14) | 46 (14) | 41 (13) | 44 (14)
RV/TLC percent predicted [Mean (Standard Deviation); unit: percent] — The RV/TLC (residual volume/total lung capacity) is a pulmonary function measure. It is an indication of air-trapping in the lungs. In general, a value over 120 percent predicted indicates that there is significant air-trapping.
  percent | 165 (27) | 158 (24) | 161 (24) | 161 (25)

OUTCOME MEASURES:

1. Primary Outcome: Exercise Endurance
Description: Exercise endurance on a constant workrate treadmill test was measured at 14 weeks. The workload on the constant workrate treadmill test corresponded to the grade and speed that the participate had reached on a symptom-limited treadmill test when they reached 85% of their peak oxygen uptake value.
Time Frame: 14 weeks
Population: We used an intent-to treat analysis using the last value carried forward. All participants were included in the final analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Breathing Retraining | Heliox | Exercise
Number analyzed (Participants) | 35 | 33 | 35
minutes | 18.1 (13.4) | 14.5 (10.7) | 11.5 (7.0)
Statistical Analysis 1: Comparison: Breathing Retraining vs Heliox vs Exercise; Test type: Superiority or Other; p = 0.015, ANCOVA — Statistical tests were 2-sided and a p value of < 0.05 was the criterion for statistical significance; The baseline value was the co-variate in this analysis

2. Secondary Outcome: Inspiratory Capacity
Description: Inspiratory capacity measured during exercise is a measure of air-trapping (dynamic hyperinflation). Inspiratory capacity was measured at an isotime (same time) during the constant workrate treadmill test at baseline and 14 weeks.
Time Frame: 14 weeks
Population: Intent-to-treat analysis was used so data on all randomized patients were analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Breathing Retraining | Heliox | Exercise
Number analyzed (Participants) | 35 | 33 | 35
Liters | 2.4 (0.7) | 2.0 (0.6) | 2.1 (0.7)
Statistical Analysis 1: Comparison: Breathing Retraining vs Heliox vs Exercise; Test type: Superiority or Other; p < 0.05, ANCOVA; The baseline value was the co-variate in this analysis

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the time period that the patient was enrolled in the study. When the patient completed the study (after 14 week testing was completed), we stopped collecting adverse event information.
Arm/Group | Breathing Retraining | Heliox | Exercise
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/33 | 5/35
Other Adverse Events (participants affected / at risk) | 1/35 | 2/33 | 1/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Breathing Retraining (N=35) | Heliox (N=33) | Exercise (N=35)
Cardiac Event (Cardiac disorders) | 1 | 0 | 3 — Patients had chest pain or needed an intervention such as angioplasty.
lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — A patient developed lung cancer during the study.
intracerebral bleed (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Patient had a intercerebral bleed during the course of the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Breathing Retraining (N=35) | Heliox (N=33) | Exercise (N=35)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) — Exacerbation of COPD that lasted over 2 weeks and caused the patient to be withdrawn from the study.
cellulitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Patient developed a cellulitis in his legs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes